CLINICAL TRIAL: NCT00634036
Title: A Randomized, Placebo-Controlled Pilot Study of Pioglitazone for the Treatment of Moderate to Severe Asthma in Obese Asthmatics
Brief Title: Pilot Study of Pioglitazone for the Treatment of Moderate to Severe Asthma in Obese Asthmatics
Acronym: GLITZ Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fernando Holguin (Other)
Collaborators: Takeda (Industry); University of Vermont (Other)
Responsible Party: Sponsor-Investigator, Fernando Holguin, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLITZ 001; 00001949
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Results first posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: Asthma; obesity; exacerbation; asthmatics; fat; overweight; adipose tissue; leptin; adiponectin; pioglitazone; Actos; wheezing; Pittsburgh; Pennsylvania; pulmonary; lung
MeSH Terms: conditions — Asthma; Obesity; Platelet Glycoprotein IV Deficiency; Overweight; Respiratory Sounds | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: pioglitazone
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pioglitazone — pioglitazone tablets: 30 mg/day for 2 weeks; then increased to 45 mg/day until week 12 (approximately 3 months)
  Other Names: Actos
  Arms: 1
Drug: placebo — matching placebo (inert tablet)
  Arms: 2

SUMMARY:
Asthmatics who are significantly overweight tend to have more severe symptoms, more flare ups, and are more likely to have poorly-controlled asthma when compared to other asthmatics.

Researchers believe this occurs because excess adipose tissue (fat) in the body can cause higher-than-normal levels of leptin and lower-than-normal levels of adiponectin in the blood.

The researchers of this study are testing a medication called pioglitazone in overweight asthmatics because they believe it can help regulate leptin and adiponectin and that this may improve symptoms of asthma.

DETAILED DESCRIPTION:
Participants in this study will be randomly assigned (like the flip of a coin) to pioglitazone or a placebo (an inactive pill). They will be given study medication to take everyday for 12 weeks (3 months).

Participants will complete a number of asthma-related questionnaires and a variety of pulmonary function tests. Participants will undergo physical exams, an electrocardiogram, and blood sampling to measure leptin, adiponectin, markers of inflammation, blood cell counts, glucose levels, BNP hormone levels, and liver function.

To monitor participants throughout the study, follow-up visits will be done at 2, 6, and 12 weeks after starting study drug. At these visits many of the pulmonary function tests and questionnaires will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosed by a physician at least 1 year prior to study enrollment
* Poorly-controlled asthma at study enrollment
* Non smokers (stopped smoking at least 1 year ago) and limited life-time history of smoking
* Body mass index 30-60
* Responds to methacholine challenge test with PC20 of <16 mg/ml
* On a stable dose of inhaled corticosteroid for at least 4 weeks prior to study entry
* FEV1 >60% predicted
* Able to obtain weekly weights at home

Exclusion Criteria:

* Systemic steroids within the past 4 weeks
* Lung pathology other than asthma
* Other significant non-pulmonary co-morbidities such as: coronary artery disease, peripheral vascular disease, cerebrovascular disease, congestive heart failure with an ejection fraction <50%, liver disease or elevated liver enzymes at baseline, malignancy (excluding non-melanoma skin cancers), AIDS, renal failure with serum creatinine >3.0, or disorders requiring steroid treatment such as vasculitis, lupus, rheumatoid arthritis
* B-type natriuretic peptide (BNP) >400 pg/mL
* Pregnant or lactating
* Currently taking a beta blocker, a CYP2C8 inhibitor or inducer such as gemfibrozil or rifampin, a TZD (thiazolidinedione), or allergic to TZD
* Taking antioxidants or nutritional supplements (stable dose of calcium, vitamin D, or multivitamin is OK)
* Illicit drug use within the past year
* Current/active upper respiratory infection (if active URI, wait until asymptomatic for 1 week to enroll)
* Asthma exacerbation within the past 4 weeks (includes ER, urgent care, or hospital visits due to asthma resulting in an increase in asthma-related medications)
* Undergoing evaluation for sleep apnea, or plans to institute treatment for sleep apnea (patients on a stable treatment regimen for sleep apnea for the last 3 months will be allowed to participate)
* Clinically significant abnormalities present on screening 12-lead electrocardiogram
* Women of childbearing potential using oral contraceptives who are not willing to use a second method of contraception during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2009-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Holguin, MD, MPH, Principal Investigator — University of Pittsburgh; Anne E. Dixon, MD, Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Vermont, Colchester, Vermont

REFERENCES:
- [Background] Hashimoto Y, Nakahara K. Improvement of asthma after administration of pioglitazone. Diabetes Care. 2002 Feb;25(2):401. doi: 10.2337/diacare.25.2.401. No abstract available. PMID 11815521
- [Background] Lee KS, Kim SR, Park SJ, Park HS, Min KH, Jin SM, Lee MK, Kim UH, Lee YC. Peroxisome proliferator activated receptor-gamma modulates reactive oxygen species generation and activation of nuclear factor-kappaB and hypoxia-inducible factor 1alpha in allergic airway disease of mice. J Allergy Clin Immunol. 2006 Jul;118(1):120-7. doi: 10.1016/j.jaci.2006.03.021. Epub 2006 May 19. PMID 16815147
- [Derived] Dixon AE, Subramanian M, DeSarno M, Black K, Lane L, Holguin F. A pilot randomized controlled trial of pioglitazone for the treatment of poorly controlled asthma in obesity. Respir Res. 2015 Nov 26;16:143. doi: 10.1186/s12931-015-0303-6. PMID 26610598
- See also: Asthma informational website — http://www.nhlbi.nih.gov/health/dci/Diseases/Asthma/Asthma_WhatIs.html
- See also: Asthma informational website — http://www.ginasthma.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pioglitazone | Placebo
Started | 12 | 11
Completed | 10 | 9
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Placebo | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (10) | 41 (14.1) | 40.2 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23
Age asthma onset [Mean (Standard Deviation); unit: years] | 15 (11) | 21 (18.9) | 18 (14.95)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 38.8 (6.8) | 43.5 (7.8) | 41.15 (7.3)
Seasonal allergies [Number; unit: participants]
  Reported allergies | 10 | 10 | 20
  Non-allergic | 2 | 1 | 3
Gastroesophageal Reflux Disease (GERD) [Number; unit: participants]
  Participants with GERD | 7 | 5 | 12
  Participants without GERD | 5 | 6 | 11
Depression [Number; unit: participants]
  Participants reporting Depression | 7 | 6 | 13
  Participants without Depression | 5 | 5 | 10
Asthma exacerbation in last 12 months [Number; unit: participants]
  Reported an exacerbation | 6 | 7 | 13
  No reported exacerbation | 6 | 4 | 10
Oral steroids in last 12 months [Number; unit: participants]
  Used oral steroids | 7 | 4 | 11
  Did not use oral steroids | 5 | 7 | 12
Inhaled corticosteroid [Number; unit: participants]
  High dose | 4 | 5 | 9
  Medium dose | 8 | 4 | 12
  Low dose | 0 | 2 | 2
Long acting beta agonist [Number; unit: participants]
  Used long acting beta agonist | 10 | 9 | 19
  Did not use long acting beta agonist | 2 | 2 | 4
Short acting beta agonist [Number; unit: participants]
  Used short acting beta agonist | 11 | 11 | 22
  Did not use short acting beta agonist | 1 | 0 | 1
Exhaled Nitric Oxide [Mean (Standard Deviation); unit: ppb] | 27.6 (27.8) | 30.8 (28.4) | 29.2 (28.1)
Immunoglobulin E [Mean (Standard Deviation); unit: IU/ml] | 291.2 (313.2) | 575 (544.7) | 433.1 (428.95)
Juniper Asthma Control [Mean (Standard Deviation); unit: scores on a scale] — Scale Range: minimum 1.0; maximum 6.0 Higher values represent increased asthma symptoms A score greater than 1.5 is considered compatible with uncontrolled asthma
  scores on a scale | 1.75 (.63) | 2.48 (1.3) | 2.115 (.965)
FEV1 (% predicted before bronchodilator use) [Mean (Standard Deviation); unit: % predicted] | 82.3 (12.1) | 81.5 (15.2) | 81.9 (13.65)
FVC (% predicted before bronchodilator use) [Mean (Standard Deviation); unit: % predicted] | 86.8 (13.7) | 85.3 (16.2) | 86.05 (14.95)
FEV1/FVC (% predicted before bronchodilator use) [Mean (Standard Deviation); unit: % predicted] | 95.3 (11.2) | 94.9 (11.12) | 95.1 (11.16)
FEV1 (% predicted after bronchodilator use) [Mean (Standard Deviation); unit: % predicted] | 77.3 (25.1) | 88.1 (4.6) | 82.7 (14.85)
FVC (% predicted after bronchodilator use) [Mean (Standard Deviation); unit: % predicted] | 79.5 (27.6) | 88.3 (16.3) | 83.9 (21.95)
FEV1/FVC (% predicted after bronchodilator use) [Mean (Standard Deviation); unit: % predicted] | 90.9 (31.2) | 97.8 (7.82) | 94.35 (19.51)

OUTCOME MEASURES:

1. Primary Outcome: Airway Reactivity
Description: Presence and degree of airway hyperresponsiveness assessed by methacholine challenge test. PC20= Methacholine dose at wich the FEV1 deops by > 20% from pre-methacholine baseline values.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: mg/ml
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 10 | 9
mg/ml | 5.08 [0 to 7.42] | 2.37 [0 to 11.22]

2. Secondary Outcome: FEV1 % Predicted
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: % predicted
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 10 | 9
% predicted | 80.3 (15) | 85.2 (12)

3. Secondary Outcome: Juniper Asthma Control Questionnaire
Description: The Juniper Asthma Control Questionnaire is a validated scale ranging from 0 to 6. Higher scores represent poorer asthma control. Values > 1.5 are compatible with poorly controlled asthma
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 10 | 9
Scores on a scale | 1.62 (.6) | 1.82 (1)

4. Secondary Outcome: Exhaled Nitric Oxide Ppb
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: ppb
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 10 | 9
ppb | 27.6 (27.8) | 30.8 (28.4)

ADVERSE EVENTS:
Arm/Group | Pioglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 12/12 | 11/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (N=12) | Placebo (N=11)
Headache (General disorders) | 7 | 4
Dizziness (General disorders) | 1 | 3
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Sore Throat (General disorders) | 5 | 2
Abdominal pain (General disorders) | 3 | 5
Nausea (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 4
Skin rash (Skin and subcutaneous tissue disorders) | 1 | 1
Muscle aches (General disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes